CLINICAL TRIAL: NCT02439307
Title: Effect of Rifaximin on Minimal Hepatic Encephalopathy and Small Intestinal Bacterial Overgrowth in Patients With Cirrhosis
Brief Title: Effycacy of Rifaximin on Reverse Minimal Hepatic Encephalopathy and Elimation Small Intestinal Bacterial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of the reconversion of the hospital to care for patients with COVID19. For this reason, it was not possible to continue recruiting and monitoring patients for this clinical study.
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Segundo Moran Villota, Titular B, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F-CNIC-2013-55
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Small Intestinal Bacterial Overgrowth; Liver Cirrhosis
Keywords: Rifaximin; Minimal hepatic encephalopathy
MeSH Terms: conditions — Liver Cirrhosis | interventions — Rifaximin; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin (Active Comparator): Patients will receive per day 1200 mg of rifaximin
  Interventions: Drug: Rifaximin
- Placebo (Placebo Comparator): Patients will receive a placebo of rifaximin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — 1200 mg of rifaximin for 2 weeks.
  Other Names: Antibiotic
  Arms: Rifaximin
Drug: Placebo — Placebo for 2 weeks
  Other Names: Action lacks substance
  Arms: Placebo

SUMMARY:
A total of 46 patients diagnosed with liver cirrhosis will be recruited. All patients will be evaluated with five psychometric tests and critical flicker frequency to diagnosis minimal hepatic encephalopathy (MHE). A breath test sample will be performed in all patients with MHE with 10 g of lactulose to establish the diagnosis of small intestinal bacterial overgrowth (SIBO). Patients diagnosed with EHM and SIBO will be randomized to receive per day 1200 mg of rifaximin (group A) or placebo (group B) for 2 weeks. A complete medical history, nutritional assessment, biochemical studies, and evaluation of quality of life will be performed in all patients included in the study. Besides the initial visit, patients will receive subsequent care 2, 4, 8, 12, and 24 weeks after the beginning of the study.

DETAILED DESCRIPTION:
MHE impairs the quality of life, increases the risk of motor vehicle accidents, and mortality. Currently, there is no consensus on treatment and yet there are few proven treatment options. Among the factors associated with MHE, is the small intestinal bacterial overgrowth (SIBO) present in 38.6% of patients with MHE. Rifaximin is a broad spectrum antimicrobial administered orally, with low risk of inducing bacterial resistance, and has been used in the treatment of MHE. It is unknown if the beneficial effect on MHE is associated with the elimination of SIBO and its efficacy when administered in patients with simultaneous diagnosis of MHE and SIBO was never been evaluated. The aim of our study is to evaluate the effect of rifaximin on MHE and SIBO in patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis of any etiology
* Men and women between 18 and 70 years.
* Patients diagnosed with minimal hepatic encephalopathy and small intestinal bacterial overgrowth
* Right-holders of the Mexican Social Security Institute
* Patients who agree to participate in the study and signed the informed consent

Exclusion Criteria:

* Recent history of alcohol abuse and/or drugs (less than 6 weeks).
* Illiterate
* Alcoholic cirrhosis
* History and/or diagnosis of overt hepatic encephalopathy
* Consumption of psychotropic medications (benzodiazepines, antiepileptics)
* Patients under treatment with lactulose, lacitol, rifaximin, neomycin, metronidazole and/or fiber supplements.
* History of chronic renal disease or heart failure
* Patients with gastrointestinal bleeding
* History of neurological or psychiatric disorders that affect the ability to develop neuropsychological tests
* Patients with diarrhea
* Diagnosis of liver cancer
* Patients with ophthalmologic disorders
* Patients taking antibiotics 30 days before the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Reversal of small intestinal bacterial overgrowth | 2 weeks
  Analyze the number of patients who reverts the small intestinal bacterial overgrowth after the study

SECONDARY OUTCOMES:
Quality of life improvement | 2 weeks
  Analyze the number of patients who improve the record of quality of life, that will be evaluated with the Chronic Liver Disease Questionnaire
Reversal of minimal hepatic encephalopathy | 2 weeks
  Analyze the number of patients who reverts the minimal hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Segundo Moran, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Centro Médico Nacional Siglo XXI, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No